CLINICAL TRIAL: NCT00784433
Title: Cardiovascular and Metabolic Effects of Moderate Alcohol Consumption in Type 2 Diabetes
Brief Title: The CArdiovasCulAr Diabetes & Ethanol (CASCADE) Trial
Acronym: CASCADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Iris Shai, Iris Shai, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOR478108CTIL
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2009-08

CONDITIONS: Diabetes; Prediabetes
Keywords: alcohol diabetes CVD
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- alcohol 1 (Experimental)
  Interventions: Dietary Supplement: alcohol
- alcohol 2 (Experimental)
  Interventions: Dietary Supplement: alcohol
- control (Placebo Comparator)
  Interventions: Dietary Supplement: alcohol

INTERVENTIONS:
Dietary Supplement: alcohol — 150 cc

SUMMARY:
Moderate alcohol may be beneficial for diabetics

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes
* Male or female alcohol abstainers (not more than 1 drink/week)
* Age between 40-75 yrs
* Clinically stable, with no history of stroke or myocardial infarction or major surgery within the previous 3 months

Exclusion Criteria:

* The use of RI or short-acting analog insulin/ pump therapy. Patients on 1-2 injections per day of NPH or long-acting analogs will be eligible for inclusion
* Triglycerides > 500 mg/dL
* HbA1c<7 or > 10%
* Serum creatinine > 2 mg/dl
* Liver dysfunction (greater than 2-fold elevation of ALT or and 3-fold elevation of AST)
* Evidence of severe diabetes complications (such as proliferative retinopathy or overt nephropathy)
* Autonomic neuropathy manifested as postural hypotension or hypoglycemia unawareness
* Patients with chronic hepatitis (C,B)
* Use of drugs that might significantly interact with alcohol such as sedatives, antihistamines, and anti-coagulants
* Presence of active cancer, or chemotherapy within the past 3 years
* Major illness that may require hospitalization
* A high potential of addictive behavior based on physician's assessment or personal or family history of addiction, alcoholism, or alcohol abuse
* Pregnant or lactating woman
* Participation in another trial with active intervention

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 6 months

SECONDARY OUTCOMES:
CVD status | 6 months

REFERENCES:
- [Derived] Golan R, Shelef I, Shemesh E, Henkin Y, Schwarzfuchs D, Gepner Y, Harman-Boehm I, Witkow S, Friger M, Chassidim Y, Liberty IF, Sarusi B, Serfaty D, Bril N, Rein M, Cohen N, Ben-Avraham S, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Stampfer MJ, Rudich A, Shai I. Effects of initiating moderate wine intake on abdominal adipose tissue in adults with type 2 diabetes: a 2-year randomized controlled trial. Public Health Nutr. 2017 Feb;20(3):549-555. doi: 10.1017/S1368980016002597. Epub 2016 Oct 3. PMID 27692023
- [Derived] Gepner Y, Golan R, Harman-Boehm I, Henkin Y, Schwarzfuchs D, Shelef I, Durst R, Kovsan J, Bolotin A, Leitersdorf E, Shpitzen S, Balag S, Shemesh E, Witkow S, Tangi-Rosental O, Chassidim Y, Liberty IF, Sarusi B, Ben-Avraham S, Helander A, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Rudich A, Stampfer MJ, Shai I. Effects of Initiating Moderate Alcohol Intake on Cardiometabolic Risk in Adults With Type 2 Diabetes: A 2-Year Randomized, Controlled Trial. Ann Intern Med. 2015 Oct 20;163(8):569-79. doi: 10.7326/M14-1650. Epub 2015 Oct 13. PMID 26458258
- [Derived] Gepner Y, Henkin Y, Schwarzfuchs D, Golan R, Durst R, Shelef I, Harman-Boehm I, Spitzen S, Witkow S, Novack L, Friger M, Tangi-Rosental O, Sefarty D, Bril N, Rein M, Cohen N, Chassidim Y, Sarusi B, Wolak T, Stampfer MJ, Rudich A, Shai I. Differential Effect of Initiating Moderate Red Wine Consumption on 24-h Blood Pressure by Alcohol Dehydrogenase Genotypes: Randomized Trial in Type 2 Diabetes. Am J Hypertens. 2016 Apr;29(4):476-83. doi: 10.1093/ajh/hpv126. Epub 2015 Aug 1. PMID 26232779